CLINICAL TRIAL: NCT05258578
Title: Telephone-Based Cognitive Behavioural Therapy for Post-Operative Bariatric Surgery Patients to Manage COVID-19 Pandemic Related Mental Health and Distress (TELE-BARICARE): A Randomized Controlled Trial to Determine Effectiveness and Adaptation for Marginalized Populations
Brief Title: Tele-BARICARE to Manage COVID-19-Related Distress
Acronym: TELE-BARICARE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Health Network, Toronto (Other)
Collaborators: Centre for Addiction and Mental Health (Other); Toronto Metropolitan University (Other); The Ottawa Hospital (Other); Humber River Hospital (Other); Thunder Bay Regional Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-5145
Record Dates: First submitted 2022-02-24; First posted 2022-02-28 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-05

CONDITIONS: Obesity; Bariatric Surgery Candidate; Mental Health Disorder; Eating Disorders
Keywords: Obesity; Bariatric Surgery; Mental Health; Disordered Eating; Cognitive Behavioural Therapy; Telephone Therapy
MeSH Terms: conditions — Obesity; Mental Disorders; Feeding and Eating Disorders; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: This study will be conducted in two parallel phases. Phase 1 is a multisite randomized controlled trial (RCT) to examine the efficacy of Tele-CBT vs. a control intervention in postoperative bariatric patients experiencing disordered eating and/or psychological distress. Qualitative exit interviews will also be conducted and data used to inform future adaptations of the intervention to meet patients' diverse needs during and post-pandemic. Phase 2 will consist of integrated knowledge translation and the creation of a diverse advisory committee to co-produce knowledge products and inform adaptation of Tele-CBT for diverse populations.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tele-CBT Group (Experimental): Participants will receive 6 weekly Tele-CBT sessions and 1 final "booster" session 1 month later, all approximately 55-minutes in duration. Briefly, the Tele-CBT sessions focus on introducing the cognitive behavioural model of overeating and obesity, scheduling healthy meals and snacks, scheduling pleasurable alternative activities to overeating, identifying and planning for difficult eating scenarios, and problem solving and challenging negative thoughts. Participants are encouraged to complete CBT homework between sessions (i.e., completing food records, pleasurable activities and worksheets). Five clinical psychology graduate students will work as study therapists under the supervision of Drs. Cassin and Sockalingam and will have biweekly case supervision meetings.
  Interventions: Behavioral: Tele-CBT
- Self-Help Resources Group (Active Comparator): Participants will be directed to the CAMH COVID-19 Self-Help webpage (www.camh.ca/covid19) to access coping tools to help with COVID-19 associated stress and anxiety, loss, grief and healing, stigma, and physical isolation. Participants in the control arm will receive weekly check-in/reminder emails for the duration of the intervention period.
  Interventions: Other: Self-Help Resources

INTERVENTIONS:
Behavioral: Tele-CBT — The Tele-CBT sessions focus on introducing the cognitive behavioural model of overeating and obesity, scheduling healthy meals and snacks, scheduling pleasurable alternative activities to overeating, identifying and planning for difficult eating scenarios, and problem solving and challenging negative thoughts. Participants are encouraged to complete CBT homework between sessions (i.e., completing food records, pleasurable activities and worksheets).
  Arms: Tele-CBT Group
Other: Self-Help Resources — Participants will be directed to the CAMH COVID-19 Self-Help webpage (www.camh.ca/covid19) to access coping tools to help with COVID-19 associated stress and anxiety, loss, grief and healing, stigma, and physical isolation.
  Arms: Self-Help Resources Group

SUMMARY:
Background: Over 60% of Canadians are overweight or obese and more than half have a history of a mental illness. The COVID-19 pandemic has made it difficult for people living with obesity to manage their weight even after undergoing bariatric surgery. These difficulties in combination with the stress of the pandemic can cause significant declines in mental health and well-being. Psychotherapy ("talk therapy") has been shown to be effective in helping to reduce mental health and disordered eating symptoms in patients managing obesity; however, there is limited data in the context of COVID-19.

Objective: This study will examine whether providing a convenient and accessible telephone-based psychotherapy during and potentially after the COVID-19 pandemic will lead to better mental health and disordered eating-related outcomes in patients managing obesity after weight loss surgery.

Hypothesis: Relative to the control group, those receiving psychotherapy will have lower mental health distress and eating disorder symptoms.

Methods: Participants recruited from 4 weight loss surgery programs across Ontario will be randomly assigned to one of two groups: 1) Control (7 weekly non-structured check-in emails and access to online COVID-19 related mental health resources) or 2) Tele-CBT (a 7-session telephone-based cognitive behavioural therapy [a type of "talk therapy"] intervention focused on developing coping skills and specifically designed for weight loss surgery patients). Participants will complete measures of mental health distress, eating behaviours and a psychological distress scale prior to and immediately following the intervention.

Implications: If Tele-CBT is found to improve post-pandemic mental health distress and eating behaviours, it could be routinely offered to patients with other chronic medical conditions as a resource to help manage psychological distress and mental health concerns emerging during and after the COVID-19 pandemic.

DETAILED DESCRIPTION:
Background: High-risk patient populations, such as those with chronic or pre-existing medical conditions, including obesity, have experienced worsening mental health, distress and eating behaviours as a result of COVID-19. Given that 63% of Canadians are classified as overweight or obese, the mental health distress associated with COVID-19 has the potential to adversely impact obesity outcomes, such as weight loss and quality of life, in patients living with obesity or undergoing bariatric surgery. Preliminary evidence for virtual mental health interventions during COVID-19 has not identified any interventions that specifically addressed psychological distress or disordered eating in patients with obesity. This is a concern given significant shifts from in-person to virtual multidisciplinary visits across obesity and bariatric programs during the pandemic.

Purpose and Research Plan: The purpose of the proposed research is to develop a virtual evidence-based treatment to improve disordered eating and psychological distress secondary to COVID-19 among diverse patients who are managing obesity after bariatric surgery. This study will be conducted in two parallel phases. Phase 1 is a multisite randomized controlled trial (RCT) to examine the efficacy of Tele-CBT vs. a control intervention in postoperative bariatric patients experiencing disordered eating and/or psychological distress. Qualitative exit interviews will also be conducted and data used to inform future adaptations of the intervention to meet patients' diverse needs during and post-pandemic. Phase 2 will consist of integrated knowledge translation and the creation of a diverse advisory committee to co-produce knowledge products and inform adaptation of Tele-CBT for diverse populations.

Impact of Research: Given the increase in mental health distress and obesogenic behaviours related to the COVID-19 pandemic, it is critical that patients have consistent access to psychosocial care. Building off our previous research, this study aims to demonstrate that Tele-CBT is an efficacious intervention for those experiencing distress secondary to the COVID-19 pandemic and to mitigate pandemic-related deteriorations in mental health, disordered eating, and weight management in obesity care. Moreover, by understanding how virtually/remotely delivered psychological interventions during COVID-19 are received and affect diverse patient populations, our study findings will inform the development and application of psychosocial treatments and services during COVID-19 and its recovery phase. Through our advisory committee, key stakeholders, and community partnerships, the investigators will disseminate our findings widely and create a plan to implement virtual psychosocial interventions in obesity care to meet the mental health needs likely to persist post-pandemic.

ELIGIBILITY:
Inclusion Criteria:

* post-operative adult bariatric patients (men, women and gender diverse individuals)
* fluent in English
* have internet access to complete online questionnaires
* meet a threshold of ≥ 5 on the Patient Health Questionnaire 9-Item scale (PHQ-9)24, a measure of depressive symptoms, or ≥ 18 on the Binge Eating Scale (BES)26, a common measure of dysregulated eating in this patient population

Exclusion Criteria:

* current active suicidal ideation
* current poorly controlled medical illness or psychiatric illness that would render Tele-CBT very difficult (e.g., psychotic disorder, bipolar disorder)
* active COVID-19 infection as it may cause neuropsychiatric symptoms that impact treatment engagement and confound study outcomes

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2022-10-06 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Change in Binge Eating Scale | Baseline (pre-intervention, when participants are enrolled), post-intervention (approximately 3-months after patients complete baseline assessment), and 3-month follow-up (approximately 6 months after patients complete baseline assessment)
  The investigators will assess change in Binge Eating Scale (BES) scores at post-intervention and at 3-month follow-up compared to baseline. The BES is a 16-item self-report measure designed specifically for use with individuals with obesity and assesses the presence of binge eating characteristics indicative of an eating disorder. Scores on the BES range from 0 to 46 with moderate and severe levels of binge eating corresponding to cut-off scores of 18 and 27, respectively.
Change in Patient Health Questionnaire-9 Item Scale | Baseline (pre-intervention, when participants are enrolled), post-intervention (approximately 3-months after patients complete baseline assessment), and 3-month follow-up (approximately 6 months after patients complete baseline assessment)
  The investigators will assess change in Patient Health Questionnaire-9 Item Scale (PHQ-9) scores at post-intervention and at 3-month follow-up compared to baseline. The PHQ-9 consists of 9-items assessing depressive symptoms on a scale ranging from 0 (not at all) to 3 (nearly every day). Scores on the PHQ-9 range from 0 to 27 with mild, moderate, moderately severe and severe levels of depressive symptoms corresponding to cut-off scores of 5, 10, 15 and 20, respectively.

SECONDARY OUTCOMES:
Emotional Eating Scale | Baseline (pre-intervention, when participants are enrolled), post-intervention (approximately 3-months after patients complete baseline assessment), and 3-month follow-up (approximately 6 months after patients complete baseline assessment)
  The investigators will assess change in Emotional Eating Scale (EES) scores at post-intervention and at 3-month follow-up compared to baseline. The EES is a 25-item self-report measure that assesses a person's tendency to cope with negative affect through eating. The scale ranges from 0 (no desire) to 4 (overwhelming urge) and consists of questions that ask participants to rate the intensity of their urge to eat in response to 25 emotions. The EES is comprised of 3 subscales that reflect eating in response to anger/frustration, anxiety, and depression.
Change in Generalized Anxiety Disorder-7 Item Scale | Baseline (pre-intervention, when participants are enrolled), post-intervention (approximately 3-months after patients complete baseline assessment), and 3-month follow-up (approximately 6 months after patients complete baseline assessment)
  The investigators will assess change in Generalized Anxiety Disorder-7 Item Scale (GAD-7) scores at post-intervention and at 3-month follow-up compared to baseline. The GAD-7 is a 7-item self-report questionnaire assessing anxiety symptoms on a scale ranging from 0 (not at all) to 3 (nearly every day). Scores on the GAD-7 range from 0 to 21 with mild, moderate and severe levels of anxiety symptoms corresponding to cut-off scores of 5, 10 and 15, respectively.
Change in Loss of Control Over Eating Scale | Baseline (pre-intervention, when participants are enrolled), post-intervention (approximately 3-months after patients complete baseline assessment), and 3-month follow-up (approximately 6 months after patients complete baseline assessment)
  The investigators will assess change in Loss of Control Over Eating Scale (LOCES) scores at post-intervention and at 3-month follow-up compared to baseline. The LOCES is a 24-item self-report measure intended to measure a global sense of loss of control overeating. Higher scores on the LOCES indicate a greater level of LOC-eating.
Kessler Psychological Distress Scale | Baseline (pre-intervention, when participants are enrolled), post-intervention (approximately 3-months after patients complete baseline assessment), and 3-month follow-up (approximately 6 months after patients complete baseline assessment)
  The investigators will assess change in Kessler (K6) scores at post-intervention and at 3-month follow-up compared to baseline. The K6 is a 6-item self-report questionnaire measuring psychological distress. Questions are scored from 0 (none of the time) to 4 (all of the time). Low scores indicate low levels of psychological distress, whereas high scores indicate high levels of psychological distress.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie E. Cassin, PhD, CPsych, Principal Investigator — Toronto Metropolitan University; Branka Agic, MD, Principal Investigator — Centre for Addiction and Mental Health Research
Locations (4):
- Canada (4):
  - The Ottawa Hospital - Civic Campus, Ottawa, Ontario
  - Thunder Bay Regional Health Sciences Centre, Thunder Bay, Ontario
  - Humber River Hospital, Toronto, Ontario
  - Toronto Western Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No
No IPD are to be shared with other researchers.

REFERENCES:
- [Derived] Sockalingam S, Leung SE, Agic B, Ma C, Hawa R, Wnuk S, Dash S, Jackson T, Akbar N, Forhan M, Cassin SE. Telephone-based cognitive behavioural therapy for patients with postoperative bariatric surgery to manage COVID-19 pandemic-related mental health issues and distress (TELE-BARICARE): a protocol for a randomised controlled trial. BMJ Open. 2022 Sep 15;12(9):e067393. doi: 10.1136/bmjopen-2022-067393. PMID 36109026